CLINICAL TRIAL: NCT05417243
Title: A Pilot Multicentre Cluster Randomised Trial to Compare the Effect of Trauma Life Support Training Programmes on Patient and Provider Outcomes
Brief Title: Effect of Trauma Life Support Training Programs on Patient Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Doctors For You (Unknown)
Responsible Party: Principal Investigator, Martin Gerdin, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tern-pilot
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Advanced Trauma Life Support (ATLS) (Experimental): Training in ATLS for residents providing trauma care.
  Interventions: Other: Trauma life support training
- Primary Trauma Care (PTC) (Experimental): Training in PTC for residents providing trauma care.
  Interventions: Other: Trauma life support training
- Standard Care (No Intervention): Trauma care according to the current standard with no intervention.

INTERVENTIONS:
Other: Trauma life support training — Clusters are randomised for their residents to be trained in one of two trauma life support training programs or to continue providing standard care.
  Arms: Advanced Trauma Life Support (ATLS); Primary Trauma Care (PTC)

SUMMARY:
Introduction:

Trauma accounts for nearly 10% of the global burden of disease. Several trauma life support programs aim to improve trauma outcomes. There is no evidence from controlled trials to show the effect of these programs on patient outcomes. We describe the protocol of a pilot study that aims to assess the feasibility of conducting a cluster randomised controlled trial comparing Advanced Trauma Life Support (ATLS) and Primary Trauma Care (PTC) with standard care.

Methods and analysis:

We will pilot a pragmatic three-armed parallel, cluster randomised, controlled trial in India, where neither of these programs are routinely taught. We will recruit tertiary hospitals and include trauma patients and residents managing these patients. Two hospitals will be randomised to ATLS, two to PTC, and two to standard care. The primary outcome will be all cause mortality at 30 days from the time of arrival to the emergency department. Our secondary outcomes will include patient, provider, and process measures. All outcomes except time to event outcomes will be measured both as final values as well as change from baseline. We will compare outcomes in three combinations of trial arms: ATLS versus PTC, ATLS versus standard care, and PTC versus standard care using absolute and relative differences along with associated confidence intervals. We will conduct subgroup analyses across the clinical subgroups men, women, blunt multisystem trauma, penetrating trauma, shock, severe traumatic brain injury, and elderly. In parallel to the pilot study we will conduct community consultations to inform the planning of the full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults (15 years or older) who present to the emergency department at participating hospitals with a history of trauma. History of trauma is here defined as having any of the external causes of morbidity and mortality listed in block V01-Y36, chapter XX of the International Classification of Disease version 10 (ICD-10) codebook as reason for presenting.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality within 30 days from the time of arrival to the emergency department | 30 days

CONTACTS AND LOCATIONS:
Locations (7):
- India (7):
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - Medica Superspecialty Hospital, Kolkata
  - Medical College, Kolkata
  - Sir Nil Ratan Sircar Medical College & Hospital, Kolkata
  - HBT Medical College And Dr. R N Cooper Municipal General Hospital, Mumbai
  - King Edward Memorial Seth G. S. Medical College and K.E.M. Hospital, Mumbai
  - Lokmanya Tilak Municipal Medical College & General Hospital, Mumbai

IPD SHARING:
Plan to Share IPD: Yes
The final anonymized dataset and code for analysis will be released publicly.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: During 2023

REFERENCES:
- [Background] Gerdin Warnberg M, Berg J, Bhandarkar P, Chatterjee A, Chatterjee S, Chintamani C, Fellander-Tsai L, Gadgil A, Ghag G, Hasselberg M, Juillard C, Khajanchi M, Kizhakke Veetil D, Kumar V, Kundu D, Mishra A, Patil P, Roy N, Roy A, David S, Singh R, Solomon H, Soni KD, Strommer L, Tandon M; Trauma life support training Effectiveness Research Network (TERN) collaborators. A pilot multicentre cluster randomised trial to compare the effect of trauma life support training programmes on patient and provider outcomes. BMJ Open. 2022 Apr 18;12(4):e057504. doi: 10.1136/bmjopen-2021-057504. PMID 35437251
- [Derived] Gerdin Warnberg M, Basak D, Berg J, Chatterjee S, Fellander-Tsai L, Ghag G, Juillard C, Khajanchi M, Khan T, Mishra A, Nandu VV, Roy N, Singh R, Soni KD, Strommer L. Feasibility of a cluster randomised trial on the effect of trauma life support training: a pilot study in India. BMJ Open. 2025 Dec 10;15(12):e099020. doi: 10.1136/bmjopen-2025-099020. PMID 41371733
- See also: Trauma life support training Effectiveness Research Network website — https://www.tern.network/